CLINICAL TRIAL: NCT05717335
Title: Observational Pilot Study With TachoSil as a Ventricular Sealant
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Tachosil-vent-2022; PI-22-078 (Registry Identifier: Ethics committee reference)
Record Dates: First submitted 2023-01-10; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Intraventricular Neoplasm
Keywords: Ventricle opening; ventricular entry; Complication; Pseudomeningocele; Cerebrospinal fluid leakage; Meningitis
MeSH Terms: conditions — Cerebral Ventricle Neoplasms; Cerebrospinal Fluid Leak; Meningitis | interventions — TachoSil; Thrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with ventricular entry during surgery (vascular, tumoral and epilepsy).: Group of patients operated on for periventricular lesions with ventricular entry and placement of TachoSil directly over the area of ventricular opening in order to avoid complications.
  Interventions: Drug: TachoSil

INTERVENTIONS:
Drug: TachoSil — Placement of TachoSil over the ventricular entry point in patients with periventricular lesions in order to avoid complications related to the ventricular entry.
  Other Names: TachoSil is a sponge sealant patch that is coated with the active substances human fibrinogen and human thrombin.

SUMMARY:
The working hypothesis in this study is that after entering the cerebral ventricular system the sealing with TachoSil is effective and safe.

A more specific hypothesis is that the use of Tachosil for brain surgery with ventricular entry reduces the number of postoperative complications (hydrocephalus, CSF leak, meningitis and pseudomeningocele).

DETAILED DESCRIPTION:
Pilot observational study with medications (MOE), single-center, prospective and retrospective study with a group of patients operated on for periventricular lesions and with ventricular entry. As it is an infrequent type of surgery in our centre, the study includes a retrospective group (same surgery and use of TachoSil).

Primary objectives:

The main objective of the study is to evaluate the effectiveness and safety of TachoSil in patients who require ventricular entry.

To evaluate the effectiveness, the percentage of complications related to the ventricular entry during surgery are recorded. These complications are hydrocephalus, CSF leak, meningitis, and pseudomeningocele.

Secondary objectives

* Intraoperative incidence of fistula after application of the ventricular patch at 20cm PEEP H20 (efficacy objective).
* Incidence of clinically confirmed percutaneous fistula during the first 30 days after surgery (efficacy objective).
* Incidence of pseudomeningocele >20cc confirmed with MRI or ultrasound (effectiveness objective).
* Incidence of radiologically confirmed hydrocephalus during the first 90 days after of the surgery.
* Record the percentage of use of other dural sealants
* Evaluate the cost effectiveness of the product.
* Describe the adverse effects related to the product
* Incidence of complication requiring reintervention within 30 days to the main surgery (safety objective).
* Assessment of the complications that are avoided: readmissions.

Study period: from December 2020 to December 2023.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for elective supratentorial surgery (tumoral, vascular or epilepsy) that during the procedure present ventricular entry, being sealed by a patch of TachoSil
* Ventricular entry during the procedure (intraoperative CSF outflow from the ventricle noticed by the surgeon)
* Adults over the age of 18
* Informed consent signed by the patient or representative (see annex 2). For cases in which the patient has died during this time a waiver of consent will be requested.

Exclusion Criteria:

* Patients or representatives who do not want to sign the consent are excluded informed, pregnant women or those under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective supratentorial craniotomy due to periventricular lesions (tumoral, vascular or epilepsy) with ventricular entry during the procedure. The TachoSil patch is used as a ventricular sealant. A part of the population will be collected prospectively and retrospective cases operated using the same systematic will also be collected.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to evaluate the effectiveness and safety of TachoSil in operated patients who require opening of the ventricle. | Up to 90 days after surgery
  To evaluate the effectiveness and the percentage of complications related to the ventricular entry during surgery. Taking into account hydrocephalus, CSF leak, meningitis and pseudomeningocele.

SECONDARY OUTCOMES:
Incidence of percutaneous CSF leakage / pseudomeningocele/ hydrocephalus/meningitis | Up to 90 days after surgery
  Percentage of complications with percutaneous CSF leakage pseudomeningocele/ hydrocephalus/meningitis

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Teixidor Rodriguez, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dasenbrock HH, Yan SC, Chavakula V, Gormley WB, Smith TR, Claus EB, Dunn IF. Unplanned Reoperation After Craniotomy for Tumor: A National Surgical Quality Improvement Program Analysis. Neurosurgery. 2017 Nov 1;81(5):761-771. doi: 10.1093/neuros/nyx089. PMID 28655201
- [Background] Eser MT, Hanalioglu S, Cetiner MZ, Dinc S, Peker HO, Sorar M, Dolgun H, Turkoglu E. Identification of Risk Factors for Postoperative Cerebrospinal Fluid Leakage and Comparison of Two Alternative Dural Augmentation Techniques in Posterior Fossa and Spinal Surgeries. Turk Neurosurg. 2019;29(3):377-385. doi: 10.5137/1019-5149.JTN.24432-18.0. PMID 30907976
- [Background] Farber H, McDowell MM, Alhourani A, Agarwal N, Friedlander RM. Duraplasty Type as a Predictor of Meningitis and Shunting After Chiari I Decompression. World Neurosurg. 2018 Oct;118:e778-e783. doi: 10.1016/j.wneu.2018.07.050. Epub 2018 Jul 17. PMID 30026145
- [Background] Grotenhuis JA. Costs of postoperative cerebrospinal fluid leakage: 1-year, retrospective analysis of 412 consecutive nontrauma cases. Surg Neurol. 2005 Dec;64(6):490-3, discussion 493-4. doi: 10.1016/j.surneu.2005.03.041. PMID 16293457
- [Result] Altaf I, Vohra AH, Shams S. Management of Cerebrospinal Fluid Leak following Posterior Cranial Fossa Surgery. Pak J Med Sci. 2016 Nov-Dec;32(6):1439-1443. doi: 10.12669/pjms.326.9956. PMID 28083041
- [Result] Behling F, Kaltenstadler M, Noell S, Schittenhelm J, Bender B, Eckert F, Tabatabai G, Tatagiba M, Skardelly M. The Prognostic Impact of Ventricular Opening in Glioblastoma Surgery: A Retrospective Single Center Analysis. World Neurosurg. 2017 Oct;106:615-624. doi: 10.1016/j.wneu.2017.07.034. Epub 2017 Jul 18. PMID 28729143
- [Result] Coucke B, Van Gerven L, De Vleeschouwer S, Van Calenbergh F, van Loon J, Theys T. The incidence of postoperative cerebrospinal fluid leakage after elective cranial surgery: a systematic review. Neurosurg Rev. 2022 Jun;45(3):1827-1845. doi: 10.1007/s10143-021-01641-y. Epub 2021 Sep 9. PMID 34499261
- [Result] Danish SF, Samdani A, Hanna A, Storm P, Sutton L. Experience with acellular human dura and bovine collagen matrix for duraplasty after posterior fossa decompression for Chiari malformations. J Neurosurg. 2006 Jan;104(1 Suppl):16-20. doi: 10.3171/ped.2006.104.1.16. PMID 16509475
- [Result] Fang C, Zhu T, Zhang P, Xia L, Sun C. Risk factors of neurosurgical site infection after craniotomy: A systematic review and meta-analysis. Am J Infect Control. 2017 Nov 1;45(11):e123-e134. doi: 10.1016/j.ajic.2017.06.009. Epub 2017 Jul 24. PMID 28751035
- [Result] Hussein K, Bitterman R, Shofty B, Paul M, Neuberger A. Management of post-neurosurgical meningitis: narrative review. Clin Microbiol Infect. 2017 Sep;23(9):621-628. doi: 10.1016/j.cmi.2017.05.013. Epub 2017 May 18. PMID 28529027
- [Result] John JK, Robin AM, Pabaney AH, Rammo RA, Schultz LR, Sadry NS, Lee IY. Complications of ventricular entry during craniotomy for brain tumor resection. J Neurosurg. 2017 Aug;127(2):426-432. doi: 10.3171/2016.7.JNS16340. Epub 2016 Nov 4. PMID 27813467
- [Result] Mistry AM, Kelly PD, Gallant JN, Mummareddy N, Mobley BC, Thompson RC, Chambless LB. Comparative Analysis of Subventricular Zone Glioblastoma Contact and Ventricular Entry During Resection in Predicting Dissemination, Hydrocephalus, and Survival. Neurosurgery. 2019 Nov 1;85(5):E924-E932. doi: 10.1093/neuros/nyz144. PMID 31058968
- [Result] Slot EMH, van Baarsen KM, Hoving EW, Zuithoff NPA, van Doormaal TPC. Cerebrospinal fluid leakage after cranial surgery in the pediatric population-a systematic review and meta-analysis. Childs Nerv Syst. 2021 May;37(5):1439-1447. doi: 10.1007/s00381-021-05036-8. Epub 2021 Feb 4. PMID 33538867
- [Result] Tu A, Tamburrini G, Steinbok P. Management of postoperative pseudomeningoceles: an international survey study. Childs Nerv Syst. 2014 Nov;30(11):1791-801. doi: 10.1007/s00381-014-2501-9. Epub 2014 Oct 9. PMID 25296539
- [Result] van Lieshout C, Slot EMH, Kinaci A, Kollen MH, Hoving EW, Frederix GWJ, van Doormaal TPC. Cerebrospinal fluid leakage costs after craniotomy and health economic assessment of incidence reduction from a hospital perspective in the Netherlands. BMJ Open. 2021 Dec 16;11(12):e052553. doi: 10.1136/bmjopen-2021-052553. PMID 34916315
- [Result] Weng J, Wu H, Wang Z. Letter to the Editor Regarding "The Prognostic Impact of Ventricular Opening in Glioblastoma Surgery: A Retrospective Single Center Analysis". World Neurosurg. 2018 Jan;109:512. doi: 10.1016/j.wneu.2017.10.067. No abstract available. PMID 29232819
- [Derived] Teixidor-Rodriguez P, Brugada-Bellsola F, Menendez-Giron S, Tardaguila-Serrano M, Gonzalez-Crespo A, Nunez-Marin F, Montane E, Busquets-Bonet J, Munoz-Narbona L, Dominguez-Alonso CJ. Effectiveness and safety of Tachosil(R) as a ventricular sealant: an observational cohort study. Acta Neurochir (Wien). 2024 Sep 27;166(1):384. doi: 10.1007/s00701-024-06276-8. PMID 39331127